CLINICAL TRIAL: NCT06187480
Title: Changes in Cardiac Functions in Patients Treated With Parathyroidectomy for Secondary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Sami Benli, Medical Doctor, Mersin University
Other Study IDs: E-78017789-050.01.04-1638902
Record Dates: First submitted 2023-12-02; First posted 2024-01-02 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Secondary Hyperparathyroidism; Myocardial Dysfunction
Keywords: Secondary hyperparathyroidism; myocardial performance index
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: underwent total parathyroidectomy
  Interventions: Procedure: total parathyroidectomy (group 1) and those who underwent subtotal parathyroidectomy (group 2)
- group 2: underwent subtotal parathyroidectomy
  Interventions: Procedure: total parathyroidectomy (group 1) and those who underwent subtotal parathyroidectomy (group 2)

INTERVENTIONS:
Procedure: total parathyroidectomy (group 1) and those who underwent subtotal parathyroidectomy (group 2) — The groups were compared according to the echocardiogram findings performed in the preoperative period and the postoperative sixth month. In addition, cardiac structure, systolic and diastolic function, especially myocardial performance index, were evaluated by echocardiography and Doppler imaging.

SUMMARY:
This study aims to investigate the changes in cardiac functions, especially myocardial performance index (MPI), in patients who underwent parathyroidectomy for secondary hyperparathyroidism.

Participants who underwent parathyroidectomy for secondary hyperparathyroidism between June 2010 and September 2021 were analyzed retrospectively. The participants were divided into two groups: those who underwent total parathyroidectomy (group 1) and those who underwent subtotal parathyroidectomy (group 2). The groups were compared according to the echocardiogram findings performed in the preoperative period and the postoperative sixth month. In addition, cardiac structure, systolic and diastolic function, especially myocardial performance index, were evaluated by echocardiography and Doppler imaging.

DETAILED DESCRIPTION:
Patient selection

The participants who developed secondary hyperparathyroidism after chronic renal failure and underwent subtotal/total parathyroidectomy in our hospital between June 2010 and September 2021 were analyzed with a single-center Nested case-control study design.

Patients with a diagnosis of chronic renal failure, secondary hyperthyroidism after chronic renal failure, preoperative and postoperative laboratory tests, parathyroidectomy operation, and preoperative and postoperative 6-month transthoracic echocardiography (ECHO) were included in the study.

Advanced-stage lung disease, atrial fibrillation, atrial and supraventricular tachycardia, extra ventricular beats, intraventricular conduction disorders, ventricular pacing, moderate to severe valve pathology, history of bypass surgery, poor image quality in transthoracic echocardiography as cardiac comorbidities Patients with disease and missing data were excluded from the study.

Data collection

Demographic data (age, gender), surgery (total/subtotal parathyroidectomy) preoperative and postoperative laboratory analyses, and ECHO reports of the patients were recorded. In laboratory values, glucose, hemoglobin, albumin, blood urea nitrogen (BUN), creatinine, calcium, phosphorus, and parathormone values were recorded. In ECHO reports, left ventricular end-diastolic diameter (cm), left ventricular end-systolic diameter (cm), left ventricular end-diastolic septum thickness (cm), left ventricular end-diastolic posterior wall thickness (cm), ejection fraction (%), fractional shortening, end-diastolic volume, end-systolic volume, ejection volume, isovolumetric relaxation time (IVRT), isovolumetric contraction time (IVCT), ejection time (ET) and myocardial performance index (MPI) data were recorded.

Surgical Technique

Patients resistant to calcimimetics and vitamin D analogs, patients with symptoms such as bone and joint pain, persistent itching, and muscle aches, and patients whose symptoms affect their quality of life are among the indications for surgery. In addition, parathyroidectomy was performed on patients with uncontrolled hyperphosphatemia, anemia hyporesponsive to erythropoietin therapy, hypercalcemia, and vascular and tissue calcifications, considered complications of SHPT.

Subtotal or total parathyroidectomy is performed in the SHPT. Total parathyroidectomy was performed without autotransplantation to prevent recurrent resistant SHPT in patients with long life expectancy and little or no possibility of kidney transplantation. In the preoperative period, routine ultrasound and 99mTc-sestamibi scintigraphy were performed on the patients. During neck exploration, tissues considered the parathyroid gland were examined as a frozen section. As a result of the frozen section, it was confirmed how many glands were removed. After parathyroidectomy was completed, intraoperative parathormone testing was performed in all patients, and it was observed that parathormone levels decreased. In the subtotal parathyroidectomy procedure, four parathyroid glands are explored. Usually, half of the parathyroid gland, closest to normal in appearance and size, is left in place with its vascular network. Other glands are excised. In the total parathyroidectomy procedure, four parathyroid glands are explored and excised. Then, a part of the parathyroid gland closest to normal in appearance and size is auto-transplanted into the sternoclaidomastoid muscle or the forearm. The transplantation area is marked with a metal clip.

Echocardiography (ECHO)

All patients were evaluated with two-dimensional, pulse-wave Doppler and tissue Doppler echocardiography. Philips HD11 XE device was used to detect echocardiographic data. Parasternal long axis view with M-Mode echocardiography method left ventricular interventricular septum thickness, left ventricular posterior wall thickness, left ventricular end-diastolic diameter, left ventricular end-systolic diameter, left ventricular end-diastolic volume, left ventricular end-systolic volume, left ventricular end-systolic volume, and fractional shortening data were determined. In addition, left ventricular stroke volume was determined by subtracting the left ventricular end-systolic volume from the left ventricular end-diastolic volume.

Myocardial performance index calculation technique

The myocardial performance index (MPI) is a numerical value obtained using cardiac time intervals. This numerical value was obtained by dividing the sum of isovolumetric contraction time (ICT) and isovolumetric relaxation time (IRT) by ejection time (ET). MPI can be detected using conventional Pulse-wave Doppler or tissue Doppler echocardiography. The mean average left ventricular (LV) MPI value is 0.39 ± 0.05. In adults, LV MPI values less than 0.40 are considered normal. Higher index values are associated with cardiac dysfunction.

Our study obtained cardiac time intervals using Pulsed wave Doppler echocardiography techniques. MPI, Pulsed wave Doppler echocardiography from the apical four-chamber images, by placing the sample volume at the endpoints of the mitral valves, the time interval between the end and the beginning of the mitral flow (a), switching to the apical five-chamber images and placing the sample volume in the left ventricular outflow tract just below the aortic valves to determine the left ventricular ET (b) was done. The left ventricular isovolumetric (ICT+IRT) sum was calculated by subtracting left ventricular ET from the time interval between the end and beginning of mitral flow (a-b). Thus, MPI [(a-b)/b] was obtained.

Statistical analysis

Mean and standard deviation were used for the statistics of continuous data. Median, minimum, and maximum values were used for continuous or ordinal data that did not show normal distribution. Frequency (n) and percentage (%) values were used to define categorical variables. Fisher's exact test was used to compare the means of two independent groups. The chi-square test was used to evaluate the relationship between categorical variables. Paired t-test was used to compare the patient's preoperative and postoperative numerical data. The statistical significance level of the data was taken as p<0.05. The statistical program www.e-picos.com was used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of chronic renal failure, secondary hyperthyroidism after chronic renal failure, preoperative and postoperative laboratory tests, parathyroidectomy operation, and preoperative and postoperative 6-month transthoracic echocardiography (ECHO) were included in the study.

Exclusion Criteria:

* Advanced-stage lung disease, atrial fibrillation, atrial and supraventricular tachycardia, extra ventricular beats, intraventricular conduction disorders, ventricular pacing, moderate to severe valve pathology, history of bypass surgery, poor image quality in transthoracic echocardiography as cardiac comorbidities Patients with disease and missing data were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients who developed secondary hyperparathyroidism after chronic renal failure and underwent subtotal/total parathyroidectomy in our hospital between June 2010 and September 2021 were analyzed with a single-center Nested case-control study design.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of myocardial performance indexes between groups | preoperatively and postoperative 6th month
  Evaluation of patients' myocardial performance indexes between groups using echocardiography and Doppler imaging in the preoperative period and at the 6th postoperative month.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University Faculty of Medicine, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benli S, Yesil E, Tazeoglu D, Ozcan C, Ozcan IT, Dag A. Changes in cardiac functions in patients treated with parathyroidectomy for secondary hyperparathyroidism. Updates Surg. 2024 Aug;76(4):1443-1452. doi: 10.1007/s13304-024-01812-8. Epub 2024 Mar 26. PMID 38530609